CLINICAL TRIAL: NCT02608502
Title: A Study to Evaluate the Efficacy of an RSV F Vaccine in Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RSV-E-301
Record Dates: First submitted 2015-11-10; First posted 2015-11-18 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Syncytial Virus (RSV)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group A (Experimental): RSV-F Vaccine (0.5mL Injection)
  Interventions: Biological: RSV-F Vaccine
- Treatment Group B (Placebo Comparator): Phosphate Buffer Placebo (0.5mL Injection)
  Interventions: Biological: Phosphate Buffer Placebo

INTERVENTIONS:
Biological: RSV-F Vaccine
  Arms: Treatment Group A
Biological: Phosphate Buffer Placebo
  Arms: Treatment Group B

SUMMARY:
The purpose of this study is to demonstrate the efficacy of the RSV F vaccine at a dose of 135µg via intramuscular (IM) injection in the prevention of moderate-severe RSV-associated lower respiratory tract disease (RSV-LRTD) in older adults ≥ 60 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥60 years of age who are ambulatory and live in the community, or in assisted-living or long-term care residential facilities that provide minimal assistance, such that the subject is primarily responsible for self-care and activities of daily living. Subjects may have one or more chronic medical diagnoses, but should be clinically stable as assessed by:

   * Absence of changes in medical therapy within one month due to treatment failure or toxicity,
   * Absence of medical events qualifying as SAEs within one month of the planned vaccination on Day 0, and
   * Absence of known, current, and life-limiting diagnoses which, in the opinion of the investigator, render survival to completion of the protocol unlikely.
2. Willing and able (on both a physical and cognitive basis) to give informed consent prior to study enrollment.
3. Able to comply with study requirements; including access to transportation for study visits.
4. Access to inbound and outbound telephone communication with caregivers and study staff.

Exclusion Criteria:

1. Participation in research involving investigational product (drug / biologic / device) within 45 days before the planned date of the Day 0 vaccination.
2. History of a serious reaction to any prior vaccination, or Guillain-Barré syndrome (GBS) within 6 weeks of any prior influenza immunization.
3. Receipt of any vaccine other than an IIV in the 4 weeks preceding the study vaccination or a pneumococcal vaccine in the 2 weeks preceding the study vaccination; or any RSV vaccine at any time.
4. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
5. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
6. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
7. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥38.0°C on the planned day of vaccine administration).
8. Known uncontrolled disorder of coagulation. Potential subjects receiving aspirin, clopidogrel, prasugrel, dipyridamole, dabigatran, apixaban, rivaroxaban or warfarin under good control for cardiovascular prophylaxis or prophylaxis of thromboembolic disease or stroke in the setting of atrial fibrillation will NOT be excluded.
9. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
10. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic, cognitive, or psychiatric conditions deemed likely to impair the quality of study compliance or safety reporting).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11850 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Numbers and percentages of subjects with moderate-severe RSV-LRTD | Day 0 to Day 182
  Defined by the presence of at least three (3) of: cough, wheezing (or worsening in baseline wheezing), new sputum production (or increase in baseline sputum production), new (or worsening) shortness of breath, and observed tachypnea (≥20 breaths per minute); plus RT-PCR-confirmed RSV infection documented within five days of symptom onset.
Numbers and percentages of subjects with solicited local and systemic AEs | Day 0 to Day 364
  Defined as solicited local and systemic AEs over the 7 days post-injection; all adverse events, solicited and unsolicited over 56 days after dosing; and MAEs, SAEs, and SNMCs over one year post dosing.

SECONDARY OUTCOMES:
Numbers and percentages of subjects with RSV-Acute Respiratory Disease (RSV-ARD) | Day 0 to Day 182
  Defined by the presence of at least one (1) of: rhinorrhea, nasal congestion, pharyngitis, cough, wheezing (or worsening in baseline wheezing), new sputum production (or increase in baseline sputum production), new (or worsening) shortness of breath; plus RT-PCR-confirmed RSV infection documented within five days of symptom onset.
RSV F protein antibody expressed as ELISA Units (EU). | Day 0 to Day 364
  Summarized by:
  * Geometric Mean Concentrations as EU (GMEU)
  * Geometric Mean Ratio (GMR)
  * Seroresponse Rate (SRR)
Palivizumab-competitive antibody (PCA) expressed as µg/mL as detected in a competitive ELISA | Day 0 to Day 364
  Summarized by:
  * Geometric Mean Concentrations as EU (GMEU)
  * Geometric Mean Fold Rise (GMFR)
Neutralizing antibody titer to at least one RSV/A and one RSV/B virus strain | Day 0 to Day 28
  Summarized by:
  * Geometric Mean Titer (GMT)
  * Geometric Mean Ratio (GMR)
Number and percentage of subjects with RSV-ARD and/or RSV-LRTD | Day 0 to Day 364
  Summarized by treatment group and by age strata and in strata defined by comorbidities and type of community housing.
Hemagglutination-inhibiting (HAI) antibody titers specific for the viruses in the 2015-16 IIV at Day 28 in the subset of subjects in each treatment group that receive IIV concurrently with study test article. | Day 0 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (60):
- United States (60):
  - Research Site US062, Birmingham, Alabama
  - Research Site US061, Mobile, Alabama
  - Research Site US046, Mesa, Arizona
  - Research Site US054, Phoenix, Arizona
  - Research Site US048, Tempe, Arizona
  - Research Site US005, Anaheim, California
  - Research Site US028, Redding, California
  - Research Site US064, San Diego, California
  - Research Site US045, Savannah, Georgia
  - Research Site US013, Stockbridge, Georgia
  - Research Site US012, Boise, Idaho
  - Research Site US069, Chicago, Illinois
  - Research Site US065, Peoria, Illinois
  - Research Site US003, Lenexa, Kansas
  - Research Site US052, Newton, Kansas
  - Research Site US058, Wichita, Kansas
  - Research Site US080, Lexington, Kentucky
  - Research Site US068, Metairie, Louisiana
  - Research Site US039, Metairie, Louisiana
  - Research Site US055, Methuen, Massachusetts
  - Research Site US072, Edina, Minnesota
  - Research Site US051, Kansas City, Missouri
  - Research Site US076, St Louis, Missouri
  - Research Site US025, Norfolk, Nebraska
  - Research Site US018, Omaha, Nebraska
  - Research Site US057, Las Vegas, Nevada
  - Research Site US059, Newington, New Hampshire
  - Research Site US066, Binghamton, New York
  - Research Site US017, Endwell, New York
  - Research Site US049, Rochester, New York
  - Research Site US078, Cary, North Carolina
  - Research Site US020, Durham, North Carolina
  - Research Site US071, Wilmington, North Carolina
  - Research Site US063, Winston-Salem, North Carolina
  - Research Site US081, Cincinnati, Ohio
  - Research Site US085, Cincinnati, Ohio
  - Research Site US030, Cleveland, Ohio
  - Research Site US053, Oklahoma City, Oklahoma
  - Research Site US044, Warwick, Rhode Island
  - Research Site US070, Charleston, South Carolina
  - Research Site US056, Mt. Pleasant, South Carolina
  - Research Site US079, Mt. Pleasant, South Carolina
  - Research Site US050, Dakota Dunes, South Dakota
  - Research Site US074, Bristol, Tennessee
  - Research Site US077, Knoxville, Tennessee
  - Research Site US029, Nashville, Tennessee
  - Research Site US047, Austin, Texas
  - Research Site US010, Dallas, Texas
  - Research Site US083, Fort Worth, Texas
  - Research Site US060, Fort Worth, Texas
  - Research Site US019, Houston, Texas
  - Research Site US084, San Angelo, Texas
  - Research Site US073, Tomball, Texas
  - Research Site US082, Salt Lake City, Utah
  - Research Site US075, Salt Lake City, Utah
  - Research Site US008, Salt Lake City, Utah
  - Research Site US027, West Jordan, Utah
  - Research Site US067, Norfolk, Virginia
  - Research Site US026, Seattle, Washington
  - Research Site US024, Marshfield, Wisconsin

REFERENCES:
- See also: Novavax Webpage — http://www.novavax.com